CLINICAL TRIAL: NCT03195231
Title: Wuling Powder for the Treatment and Underlying Mechanism of Depressive Symptoms in Patients With Parkinson's Disease: a Randomised, Double-blind, Placebo-controlled Trial.
Brief Title: Wuling Powder for the Treatment and Underlying Mechanism of Depressive Symptoms in Patients With Parkinson's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Hospital (Other Government)
Collaborators: Tongji Hospital (Other); Shanghai Tong Ren Hospital (Other); The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Wen Su, Clinical professor and Principal investigator, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 121-2016009
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Antidepressive Agents
Keywords: Parkinson's disease; Depression; Wuling Powder
MeSH Terms: conditions — Parkinson Disease; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wuling Powder Group (Experimental): Take Wuling Powder 3 times a day，3 pills each time for 12 weeks
  Interventions: Drug: Wuling Powder
- Placebo Group (Placebo Comparator): Take placebo drug which cannot be distinguished from the experimental drug 3 times a day，3 pills each time for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Wuling Powder — Patients of Wuling Group are instructed to take Wuling Powder 3 times a day and 3 pills each time for 12 weeks.
  Arms: Wuling Powder Group
Drug: Placebo — Patients of Placebo Group are instructed to take placebo drug 3 times a day and 3 pills each time for 12 weeks.
  Arms: Placebo Group

SUMMARY:
Depression is one of the most important nonmotor features of idiopathic PD（Parkinson's disease ）which may not just interfere with the motor symptoms of PD but can also cause immense personal suffering as well as decreased quality of life with increased disability and caregiver burden. However,there is little hard evidence to guide clinical treatment. Although some newer dopamine agonists also have antidepressive effect, the use of tricyclic or nontricyclic antidepressants is frequently required.However, the side-effects of these agents may also worsen some preexisting nonmotor problems in PD. Wuling powder is a Chinese medicine which is made by cultivating Xylariasp mycelium using submerged fermentation technology. Xylariasp is the fungus sclerotia which grow in termite nests. Wuling powder is mainly used to soothe nerves and anti-insomnia in clinical. The antidepressant effect of Wuling powder has been confirmed in clinical, but not in the patients of Parkinson's disease. Therefore, the investigators design a randomized, double-blind, placebo-controlled study to evaluate the antidepressant effect of Wuling powder in PD patients and its underlying mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic Parkinson's disease according to the 2015 MDS（Movement Disorder Society）-PD criterion
2. Hoehn-Yahr stage: 1-3
3. Under steady therapy of antiparkinsonian drugs for at least 28 days
4. HAMD≥13
5. MMSE（Mini-Mental State Examination）≥24
6. Neither use antidepressant drugs nor antipsychotic drugs within 4 weeks
7. Signed informed consent

Exclusion Criteria:

1. Have other psychotic symptoms
2. Suicide ideation or behavior
3. Severe cognitive impairment，chronic organs failure，malignant tumors
4. Glutamic-pyruvic transaminase or glutamic oxalacetic transaminase≥1.5 times of the high normal range or white blood cell<4*10^9/L or serum creatinine>84umol/L
5. Pregnancy or lactation period
6. Participant in other trials or have taken other experimental drugs within 90 days
7. Allergic to fungal food or fungal drugs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-06-25 (Estimated); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
the change of depression from baseline to 12 weeks | 12 weeks after treatment
  the change of depression from baseline to 12 weeks,as assessed with the use of HAMD（Hamilton Depression Scale）

CONTACTS AND LOCATIONS:
Overall Officials: Wen Su, Principal Investigator — Beijing Hospital